CLINICAL TRIAL: NCT04352946
Title: Protecting Health Care Workers From COVID-19 With Hydroxychloroquine Pre-exposure Prophylaxis: A Randomized, Placebo-controlled Trial
Brief Title: HEalth Care Worker pROphylaxis Against COVID-19: The HERO Trial
Acronym: HERO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GeoSentinel Foundation (Other)
Responsible Party: Principal Investigator, Bradley A. Connor, M.D., Clinical Professor of Medicine, Weill Cornell Medicine, GeoSentinel Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GFICOVID-19-1
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Prophylaxis; COVID-19; Health Care Worker; Hydroxychloroquine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: HCW are randomized to either the study drug (HCQ) or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in the study will be randomized to either the investigational drug (HCQ) or placebo. The investigational drug and placebo will have identical appearance and be taken at the same frequency and dosage. The administration of the drug and assessment will be blinded. Study arms will be unmasked at the end of the study for the final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrocholoroquine Pre-exposure prophylaxis (Experimental): HCQ will be administered as 400mg orally once for 60 days.
  Interventions: Drug: Hydroxychloroquine Pre-Exposure Prophylaxis
- Placebo (Placebo Comparator): Placebo will be administered as 400mg orally once for 60 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine Pre-Exposure Prophylaxis — HCQ PreP 400mg daily
  Other Names: Hydroxychloroquine PreP; HCQ PreP
  Arms: Hydrocholoroquine Pre-exposure prophylaxis
Drug: Placebo oral tablet — Placebo tablets 400mg daily
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blinded, randomized placebo-controlled trial to determine if pre-exposure prophylaxis (PrEP) with 400mg hydroxychloroquine (HCQ), taken orally once daily, for health care workers in the hospital reduces symptomatic and asymptomatic COVID-19 disease during the pandemic. 374 health care workers will be randomized at a 1:1 allocation between the intervention and placebo arms and followed for 90 days. The cumulative incidence of COVID-19 infection in the intervention group will be compared to the cumulative incidence of COVID-19 in the placebo group with relative (risk ratio and 95% CI) and absolute measures (risk difference and 95% CI).

DETAILED DESCRIPTION:
This is a double-blinded, randomized placebo-controlled trial to determine if pre-exposure prophylaxis (PrEP) with 400mg hydroxychloroquine (HCQ), taken orally once daily, for health care workers in the hospital reduces symptomatic and asymptomatic COVID-19 disease during the pandemic.

Secondary outcomes include 1) Adverse events; 2) Duration of symptomatic COVID-19 disease; 3) Days hospitalized attributed to COVID-19; 4) Respiratory failure attributable to COVID-19 disease requiring i) non-invasive ventilation or ii) intubation/mechanical ventilation; 5) Mortality attributed to COVID-19 disease, and; 6) Number of days unable to work attributed to COVID-19. Laboratory markers within participants with confirmed COVID-19 will also be explored.

A total of 374 HCW will be randomized using a fixed 1:1 allocation ratio with randomization in permuted block of varying sizes from four to eight will be used to ensure equal allocation to each group. The study population will be health care workers at the New York Presbyterian Hospital - Cornell Campus and they will participate in the study for 90 days.

To determine if the intervention has been successful, the cumulative incidence of COVID-19 infection in the intervention group will be compared to the cumulative incidence of COVID-19 in the placebo group with relative (risk ratio and 95% CI) and absolute measures (risk difference and 95% CI). Investigators will also calculate adjusted risk ratios and risk differences including job class as a covariate and any other baseline clinical and demographic characteristics that are not balanced between the treatment and placebo arms using a log-binomial regression model.

ELIGIBILITY:
Inclusion Criteria:

1. Health care worker (HCW) at the hospital who work on a "full time" basis during the study period. For the purposes of the study, "health care workers" are physicians, nurses, nurse practitioners, physician assistants, respiratory therapists, X-ray technicians, social workers and support staff (including but not limited to house-keeping, and porters).
2. Age ≥18 years.
3. Ability to communicate with study staff in English

Exclusion Criteria:

1. Known hypersensitivity/allergy to hydroxychloroquine or to 4-aminoquinoline compounds.
2. Current use of hydroxychloroquine for the treatment of a medical condition.
3. Known prolonged QT syndrome, or concomitant medications which simultaneously may prolong the QTC that cannot be temporarily suspended/replaced. These are including but not limited to Class IA, IC and III antiarrhythmics; certain antidepressants, antipsychotics, and anti-infectives; domperidone; 5-hydroxytryptamine (5-HT)3 receptor antagonists; kinase inhibitors; histone deacetylase inhibitors beta-2 adrenoceptor agonists.
4. Known pre-existing retinopathy of the eye.
5. Disclosure of self-administered use of hydroxychloroquine or chloroquine currently under investigation <4 weeks prior to study. This window is intended to account for the drug half-life of HCQ (21 days).
6. Baseline symptom of COVID-19 disease at enrollment and baseline viral detection specimen positive for SARS-COV-2. All participants with COVID-19 symptoms at enrollment will be directed to have confirmatory testing (within the department or occupational health as per the site guidelines). Participants who are negative for SARS-COV-2 will be redirected to enrollment procedures, those testing positive will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2020-04-24 (Estimated); Primary Completion 2020-06-24 (Estimated); Study Completion 2020-08-24 (Estimated)

PRIMARY OUTCOMES:
Cumulative Incidence of COVID-19 Infection | 90 days
  Incidence of symptomatic and asymptomatic COVID-19 infection in health care workers

SECONDARY OUTCOMES:
Adverse events incidence | 90 days
  Incidence of reported and grade of adverse events
Duration of symptomatic COVID-19 disease | 90 days
  Duration in days of symptomatic COVID-19 disease in HCW who had disease
Days hospitalized attributed to COVID-19 | 90 days
  Duration in days of hospitalization attributed to COVID-19 disease in HCW who had disease
Number or respiratory failure attributable to COVID-19 disease | 90 days
  Number of HCW with respiratory failure attributable to COVID-19 disease requiring i) non-invasive ventilation or ii) intubation/mechanical ventilation in HCW who developed disease
Mortality Incidence | 90 days
  Cumulative Incidence of Mortality attributed to COVID-19 disease in HCW who developed disease
Days of work lost | 90 days
  Number of days unable to work attributed to COVID-19 in HCW who developed disease

OTHER OUTCOMES:
Proportion of HCW with plasma able to neutralize SARS-CoV-2 virus | 90 days
  Proportion of participants with plasma able to neutralize SARS-CoV-2 virus (plaque reduction neutralization test) in vitro.
Number of participants with severity markers of host immune and endothelial activation | 90 days
  Number of participants with severity markers of host immune and endothelial activation measured at clinical presentation and their ability to predict severity and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley A Connor, MD, Principal Investigator — Dr. Bradley A. Connor
Locations (1):
- The New York Center for Travel and Tropical Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
supporting made available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From July 1, 2020 until December 31, 2020
Access Criteria: from our web site
URL: http://www.geosentinel.com